CLINICAL TRIAL: NCT06673381
Title: Prediction of Acute Coronary Syndrome In-hospital Major Adverse Cardiovascular Events by High Sensitivity C- Reactive Protein to Albumin Ratio
Brief Title: High Sensitive C-reactive Protein to Albumin Ratio in Acute Coronary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Elbasuony Morsy, Resident at internal medicine department, Sohag University
Other Study IDs: AEMorsy
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Acute Coronary Syndrome
Keywords: high sensitive c-reactive protein to albumin ratio
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum albumin , serum high sensitive c-reactive protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- high sensitive c-reactive protein to albumin ratio (hs-CAR): Group A ( patients with high hs-CAR) and group B ( patients with low hs-CAR)

SUMMARY:
assess the use of hs- C-reactive protein to albumin ratio (hs-CAR) in prediction of in-hospital short-term major adverse cardiac events (MACEs) in acute coronary syndrome (ACS) patients

DETAILED DESCRIPTION:
Observational study conducted at coronary care unit(CCU) in sohag university hospital It included patients with ACS diagnosed according to AHA/ACCF guidelines (according to symptoms, ECG findings and serum troponin levels), who had admitted to the CCU.

Venous blood samples were instantly collected on admission to the hospital. hs-CRP , serum albumin level were measured.

hs-CAR is calculated and the patients divided into two groups: Group A ( patients with high hs-CAR) and group B ( patients with low hs-CAR) In-hospital MACE was regarded as the end point of our study. It was defined as acute heart failure, cardiogenic shock, reinfarction, all-cause death, serious arrhythmia and cardiac death

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 Year or older presented by ACS not candidet for primary percutaneus coronary intervention ( PCI ) .

Exclusion Criteria:

* • Patients aged < 18 years old

  * Patients who have eGFR <60 ml/kg /m2
  * Patients who have malignancies
  * Patients who have chronic heart failure (NYHA class >II)
  * Pateints who have chronic liver disease
  * Patients who have nephrotic syndrome
  * Patients who have acute cerebrovascular stroke
  * Pregnant women
  * Patients who have recent infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It included patients with ACS diagnosed according to AHA/ACCF guidelines according to symptoms, ECG findings and serum troponin levels), who had admitted to the CCU.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
assess the use of hs- C-reactive protein to albumin ratio (hs-CAR) in acute coronary syndrom patients | at time of admission in hospital
  Venous blood samples were collected on admission to the hospital. hs-CRP , serum albumin level were measured.
  hs-CAR is calculated and the patients divided into two groups: Group A ( patients with high hs-CAR) and group B ( patients with low hs-CAR)

CONTACTS AND LOCATIONS:
Overall Officials: Amira Elbasuony, resident, Principal Investigator — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided